CLINICAL TRIAL: NCT04278222
Title: Efficacy and Safety of Anlotinib Plus Toripalimab as First-line Regimen in Frail Patients (ECOG 2) With Advanced Gastric Cancer (APICAL-GC): an Open-label, Single Arm, Phase II Trial
Brief Title: Anlotinib Plus Toripalimab as First-line Treatment for Advanced Gastric Cancer With ECOG 2 (APICAL-GC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Director, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APICAL-GC
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Immunotherapy; Anlotinib; Toripalimab
MeSH Terms: conditions — Stomach Neoplasms | interventions — anlotinib; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Plus Toripalimab (Experimental): the combination of Anlotinib Plus Toripalimab as first-line treatment
  Interventions: Drug: Anlotinib Plus Toripalimab

INTERVENTIONS:
Drug: Anlotinib Plus Toripalimab — Anlotinib 12mg oral administration daily d1-d14, q3w; Toripalimab 240mg iv drop d1, q3w

SUMMARY:
This study is designed to evaluate the efficacy and safety of the combination of Anlotinib wiht Toripalimab in advanced gastric cancer with ECOG 2 as first-line regimen.

DETAILED DESCRIPTION:
Anlotinib is a new, orally administered tyrosine kinase inhibitor that targets vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptors (PDGFR), and c-kit. Toripalimab is a humanized immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed cell death 1 (programmed death-1; PD-1), with potential immune checkpoint inhibitory and antineoplastic activities. In the present study, we design a single-arm, single center Phase II trial to evaluate the efficacy and safety of the combination of Anlotinib wiht Toripalimab in advanced gastric cancer with ECOG 2 as first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, UICC stage IV gastric cancer;
* no prior systematic anti-cancer treatment and relapse or metastases was occurred more than 12 months after adjuvant chemotherapy;
* at least one measurable lesion;
* received radiotherapy 3 weeks before recruitment, but the lesion undergoing radiotherapy could not be used to calculate clinical benefit using RECISET criteria;
* ECOG performance status 2;
* the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN), ALT and AST <2.5 × ULN and if liver metastases, BIL < 3 × ULN, ALT and AST <5 × ULN; Serum Cr ≤ 1.5 × ULN;
* Patient's written declaration of consent obtained;
* Estimated life expectancy > 3 months;

Exclusion Criteria:

* harboring HER2 positive including IHC 3+ or IHC 2+ with Fish positive;
* dMMR/MSI-H;
* Myocardial infarction, unstable angina pectoris, Grade III or IV heart failure (NYHA classification);
* have received anlotinib or other immune checkpoint inhibitor ;
* with known or clinically suspected brain metastases, autoimmune disease, organ transplantation ;
* severe wounds or surgery 4 weeks before recruitment;
* received glucocorticoid (more than 10mg prednisone ) and immunosuppressive agents;
* History of a second malignancy during the past 5 years before inclusion in the study or during participation in the study, with the exception of a dermal basal cell or squamous cell carcinoma or cervical carcinoma in situ, if these were treated curatively.
* pregnancy or breast feeding;
* absent or restricted legal capacity;
* a significant concomitant disease which, in the investigating physician's opinion, rules out the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 8 weeks
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission

SECONDARY OUTCOMES:
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 8 weeks
  Time from treatment beginning until disease progression
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 8 weeks
  Time from treatment beginning until death from any cause
Deepness of response | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 8 weeks
  Investigation of depth of response during first-line treatment
Disease control rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 8 weeks
  Proportion of patients with reduction and non-change in tumor burden of a predefined amount, including complete remission, partial remission and stable disease
adverse events | Through study completion, an average of 4 weeks
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Shanghai Changzheng Hospital, Shanghai, China

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069